CLINICAL TRIAL: NCT03599661
Title: Developing and Validating Fertilit-e: An eHealth Fertility Preservation Decision Aid for Young Adults With Cancer - Aim 1
Brief Title: Developing and Validating Fertilit-e
Status: Terminated | Type: Observational
Why Stopped: PI decision - competing study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00047585; CCCWFU 01717 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Malignant Neoplasm
Keywords: Cancer; Fertility; Preservation
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fertilit-e: Participants review Fertilit-e content, undergo interviews about issues of content, functionality, and ease of use, and complete questionnaires over 45-60 minutes.
  Interventions: Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Participants will review a computer prototype of Fertilit-e alpha. Using an interview guide, participants will be asked about issues of content, functionality, and ease of use (i.e., comprehensibility and usability). Interviews will be completed within 45-60 minutes.
Other: Questionnaire Administration — All participants will complete an interviewer administered screener for health literacy and self-report items for technology use, eHealth literacy, and need for cognition.

SUMMARY:
The main purpose of this project is to adapt and validate an eHealth fertility preservation decision-making support tool (Fertilit-e) for young adults with cancer.

DETAILED DESCRIPTION:
The overarching goal is to utilize innovations in eHealth technology to address fertility preservation knowledge deficits and decision-making options for young adults with cancer ages 18-39 years of age. Every year, approximately 70,000 young adults (ages 18-39) are diagnosed with cancer, which can significantly affect their health-related quality of life in multiple areas, including the potential for infertility or other reproductive challenges. Despite this, very few young adults diagnosed with cancer are actually provided fertility preservation information let alone effective strategies or tools for how to best navigate their fertility preservation options. It is critical to provide decision-making information and support about infertility risk and existing interventions to maintain reproductive potential in a delivery mode that is most congruent with this population's health communication style, such as eHealth applications.

The goal is to adapt and optimize fertility preservation content in a tailored mHealth tool for fertility preservation decision-making. More specifically, the team will adapt fertility-preservation content for tailored, rapid, and clear dissemination of information in an engaging, cross-platform, patient-friendly mHealth format. The study team will alpha-test this tool with an ethnically diverse sample of cross-cultural end users to collect qualitative data and evaluate usability and comprehensibility to refine content and design. No formal hypothesis testing will be done.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of cancer during ages 15 to 39.
* Will be receiving or have received treatment associated with a risk of infertility (i.e., systemic chemotherapy, pelvic radiotherapy, and/or pelvic surgery with potential impact on reproductive function).
* Considered or wish they had considered fertility preservation treatments.
* Able to speak, read, and understand English.
* Able to provide informed consent.
* Have internet access.
* Have a laptop or desktop computer that can connect to WebEx.

Exclusion Criteria:

* Infertility diagnosis prior to cancer diagnosis.
* History of fertility preservation or fertility treatments prior to their cancer diagnosis.
* Are more than five years post-cancer-related treatments (i.e., systemic chemotherapy, pelvic radiotherapy, and/or pelvic surgery).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults with cancer who are currently ages 18 to 39.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Salsman, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fertilit-e
Started | 21
Completed | 12
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Population: 21 participants were enrolled/consented. Nine participants were lost to follow up and no data was collected. Only 12 participants have data that was collected.
Arm/Group | Fertilit-e
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Fertilit-e Alpha - Usability (Number of Participants)
Description: To evaluate Fertilit-e alpha, we will examine its usability through a series of think aloud interviews. Qualitative analysis will provide an integrative summary and identification of key points, potential themes, and areas of further exploration.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fertilit-e
Number analyzed (Participants) | 12
Participants
  Homepage: Usable | 4
  Homepage: Not usable | 8
  Risks/Options: Usable | 6
  Risks/Options: Not usable | 6
  Personal Stories: Usable | 9
  Personal Stories: Not usable | 3
  Financial Concerns: Usable | 8
  Financial Concerns: Not usable | 4
  FAQ: Usable | 9
  FAQ: Not usable | 3
  Personal Summary: Usable | 5
  Personal Summary: Not usable | 7

2. Primary Outcome: Evaluation of Fertilit-e Alpha- Usability (System Usability Scale)
Description: To evaluate Fertilit-e alpha, we will examine its usability through the System Usability Scale, a simple, ten-item attitude Likert scale (1 - strongly disagree to 5 strongly agree) giving a global view of subjective assessments of usability. The score range is 0 to 100. Higher scores are better and scores above 68 are considered above average.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fertilit-e
Number analyzed (Participants) | 12
score on a scale | 85.0 (15.5)

3. Secondary Outcome: Evaluation of Fertilit-e Alpha- Comprehensibility
Description: To evaluate Fertilit-e alpha, we will examine its comprehensibility and design through a series of think aloud interviews. Qualitative analysis will provide an integrative summary and identification of key points, potential themes, and areas of further exploration.
Time Frame: 6 months
Population: All 12 participants for Personal Stories, FAQ, and Personal Summary did not provide data for these themes.
Measure: Count of Participants; unit: Participants
Arm/Group | Fertilit-e
Number analyzed (Participants) | 12
Participants
  Homepage: Comprehensible | 8
  Homepage: Not comprehensible | 4
  Risks/Options: Comprehensible | 9
  Risks/Options: Not comprehensible | 3
  Personal Stories: number analyzed (Participants) | 6
  Personal Stories: Comprehensible | 5
  Personal Stories: Not comprehensible | 1
  Financial Concerns: Comprehensible | 4
  Financial Concerns: Not comprehensible | 8
  FAQ: number analyzed (Participants) | 6
  FAQ: Comprehensible | 5
  FAQ: Not comprehensible | 1
  Personal Summary: number analyzed (Participants) | 0
  Personal Summary: Comprehensible | 0
  Personal Summary: Not comprehensible | 0

ADVERSE EVENTS:
Time Frame: No adverse events were collected for this study.
Description: Adverse events were not collected for this study.
Arm/Group | Fertilit-e
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT03599661/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT03599661/ICF_001.pdf